CLINICAL TRIAL: NCT00872755
Title: Laparoscopic Nissen Fundoplication Combined With Posterior Gastropexy in Surgical Treatment of Gastroesophageal Reflux Disease
Brief Title: Nissen and Gastroplasty in Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Responsible Party: Evangelos C. Tsimoyiannis, G. Hatzikosta General Hospital, Ioannina, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GH-1948-02; GHDS-12345-2
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia; Barrett's Esophagus; Esophagitis; Dysphagia
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Barrett Esophagus; Esophagitis; Deglutition Disorders | interventions — Fundoplication; Gastropexy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nissen (Active Comparator): Laparoscopic Nissen Fundoplication
  Interventions: Procedure: Nissen
- Gastropexy (Active Comparator): Procedure/Surgery Laparoscopic Nissen Fundoplication combined with posterior gastropexy
  Interventions: Procedure: Nissen; Procedure: Gastropexy

INTERVENTIONS:
Procedure: Nissen — Laparoscopic Nissen Fundoplication
Procedure: Gastropexy — posterior gastropexy
  Arms: Gastropexy

SUMMARY:
Laparoscopic Nissen Fundoplication has established itself as the procedure of choice in the surgical management of the majority of patients suffering from gastroesophageal reflux disease (GERD). Postoperative paraesophageal herniation has incidence ranges up to 7% in the immediate postoperative period. This randomized controlled study was scheduled to investigate the role of the posterior gastropexy, in combination with laparoscopic Nissen fundoplication, in prevention of paraesophageal herniation and improvement of postoperative results, in surgical treatment of GERD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Indications for surgical treatment of GERD
* ASA I, II

Exclusion Criteria:

* ASA III, IV
* Previous gastric procedures
* Conversion to open procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-01; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Laparoscopic Nissen fundoplication combined with posterior gastropexy may prevent postoperative paraesophageal or sliding herniation in surgical treatment of GERD | 9-94 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos C. Tsimoyiannis, M.D. chairman, Study Chair — G. Hatzikosta General Hospital, Ioannina, Greece
Locations (1):
- G. Hatzikosta General Hospital Department of Surgery, Ioannina, Epirus, Greece

REFERENCES:
- [Derived] Tsimogiannis KE, Pappas-Gogos GK, Benetatos N, Tsironis D, Farantos C, Tsimoyiannis EC. Laparoscopic Nissen fundoplication combined with posterior gastropexy in surgical treatment of GERD. Surg Endosc. 2010 Jun;24(6):1303-9. doi: 10.1007/s00464-009-0764-0. Epub 2009 Dec 4. PMID 19960205